CLINICAL TRIAL: NCT01381406
Title: Impact of Initiating Tiotropium Alone Versus Initiating Tiotropium in Combination With Fluticasone Propionate/Salmeterol Xinafoate Combination (FSC) on Chronic Obstructive Pulmonary Disease-related Outcomes in Patients With Pre-existing Exacerbations
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111266
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2011-10-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients: Patients who are at least 40 years of age and diagnosed with COPD using ICD-9 codes of 491.xx, 492.xx, and 496.xx in an administrative claims database.
  Interventions: Drug: TIO; Drug: TIO+FSC

INTERVENTIONS:
Drug: TIO — Patients receiving tiotropium bromide at index within the study period.
  Other Names: Spiriva®
Drug: TIO+FSC — Patients receiving tiotropium bromide plus fluticasone propionate-salmeterol xinafoate combination at time of index within the study period.
  Other Names: Spiriva ® + ADVAIR ®

SUMMARY:
This was a retrospective cohort design using administrative claims data from Jan 1, 2003 through Sep 30, 2007, representing the years of available data, were used for this study. Managed care enrollees having at least one pharmacy claim for tiotropium (TIO) during the study period were identified as the target population. An index TIO prescription was defined as the first chronologically occurring pharmacy claim for TIO during the period Jan 1, 2004 to Aug 31, 2006, called the enrollment period. The date of the index TIO prescription was termed as the index Rx date, and the 1-year period before the index Rx date was termed as the pre-index period. The period after the index date was termed as the post-index date, and is further divided into a 30-day combination assessment period and a 1-year follow-up period. COPD clinical and economic outcomes were measured in a variable length follow up period.

The combination assessment period, defined as the 30-day period following the index Rx date, was used to categorize patients into 2 cohorts: TIO alone or TIO + FSC (fluticasone propionate/salmeterol xinofoate combination) depending on whether they use FSC in combination with TIO during this period. Combination therapy with TIO + FSC was defined as having an FSC claim on the same date as the TIO claim or a TIO and FSC pharmacy claim with overlapping days supply occurring within 30 days of index Rx date. Enrollees adding FSC for the first time after the 30-day combination assessment period were excluded from the sample, thus ensuring that the TIO-alone cohort is not using FSC. No outcomes were assessed in the 30-day combination assessment period. The 1-year period after the end of the 30-day combination assessment period was termed as the follow-up period and was used to assess all study outcomes. Enrollees were required to be continuously eligible in their health plans during the pre-index and post-index periods for a total of 25 months. An intent-to-treat approach was used for the analyses. Thus, patients identified to be in a drug therapy cohort were considered to be using that therapy during the entire follow-up period, regardless of therapy discontinuations.

Specifically the study hypothesis for the primary outcome being tested was:

Ho: There is no difference in risk of any COPD-related exacerbation between TIO+FSC and TIO cohorts Ha: There is a difference in risk of any COPD-related exacerbation between TIO+FSC and TIO cohorts

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between TIO+FSC and TIO cohorts Ha: There is a difference in COPD-related costs between TIO+FSC and TIO cohorts

ELIGIBILITY:
Inclusion Criteria:

* Continuous health plan eligibility in the pre- and post-index periods
* age ≥40 years at the index date
* Presence of at least 1 claim with an ICD-9-CM code for COPD in any diagnosis field (490.xx, 491.xx, 492.xx, 496.xx) in the pre- and post-index period
* ≥1 exacerbation in the pre-index period (defined as a COPD-related Emergency Room visit or hospitalization)
* ≥1 prescription claim for ipratropium or ipratropium/albuterol combination in the pre-index period
* an index event of at least one pharmacy claim for TIO (tiotropium) combination in the pre-index period during the study period (January 1, 2003 through April 30, 2008)
* ≥2 prescriptions for TIO (including the index prescription) during the post-index period

Exclusion Criteria:

* presence of comorbid conditions (respiratory cancer, cystic fibrosis, fibrosis due to tuberculosis [TB], and bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary TB, sarcoidosis) during the pre- and post-index periods
* use of FSC in pre-index period
* exacerbation (emergency room visit or hospitalization) within 30 days after the index date

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data for managed-care enrollees age 40 and older with a diagnosis of COPD and an index event of at least one pharmacy claim for TIO during the study period (January 1, 2003 through April 30, 2008) were identified. Subjects were required to have ≥1 exacerbation in the pre-index period (defined as a COPD-related emergency room visit or hospitalization), ≥1 prescription claim for ipratropium or ipratropium/albuterol combination in the pre-index period, ≥2 prescriptions for TIO (including the index prescription) during the post-index period, no prescription for FSC during the pre-index period, and no exacerbation or hospital/emergency room visit within 30 days after the index date. ICD-9-CM code 490.xx, bronchitis not specified as chronic or acute, was included in an attempt to enhance the validity of the analysis by capturing patients with chronic bronchitis whose condition was coded incorrectly.
Sampling Method: Non-Probability Sample
Enrollment: 3333 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Pre-assignment Details: Participants were treated with tiotropium bromide (TIO) or tiotropium bromide plus fluticasone propionate/salmeterol xinafoate combination (TIO + FSC) by their practitioners, and the database included information about their healthcare encounters.
Groups:
- Tiotropium Bromide (TIO): Patients receiving tiotropium bromide (TIO) at the index date within the study period
- TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC): Patients receiving TIO plus fluticasone propionate (FSC)/salmeterol xinafoate combination (TIO + FSC) at the time of the index date within the study period
Period: Overall Study
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC)
Started | 2481 | 852
Completed | 2481 | 852
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC) | Total
Number analyzed (Participants) | 2481 | 852 | 3333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (10.9) | 64.6 (11.0) | 65.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1166 | 399 | 1565
  Male | 1315 | 453 | 1768
Number of health care encounters, as a measure of resource utilization [Number; unit: number of encounters] — The number of health care encounters for each participant group was measured. COPD = Chronic Obstructive Pulmonary Disease. An exacerbation of COPD is defined as an emergency department visit and a primary COPD diagnosis code or a physician visit plus COPD prescription (moderate) or hospitalization with a primary diagnosis of COPD (severe).
  number of encounters
    Home oxygen therapy | 801 | 248 | 1049
    Intensive care unit stays for COPD | 81 | 29 | 110
    Severe exacerbation of COPD | 360 | 175 | 535
    Moderate exacerbation of COPD | 2274 | 747 | 3021
    Hospitalization for COPD | 467 | 228 | 695
    Emergency department visit for COPD | 570 | 199 | 769
Mean number of health care encounters, as a measure of resource utilization [Mean (Standard Deviation); unit: number of encounters] — The mean number of health care encounters for each participant group was measured. COPD = Chronic Obstructive Pulmonary Disease. SABA = Short Acting Beta Agonist.
  number of encounters
    SABA containers | 2.4 (5.0) | 2.2 (5.4) | 2.4 (5.1)
    Oral corticosteriod prescriptions | 2.1 (2.9) | 1.9 (2.3) | 2.0 (2.8)
    Number of physician visits for COPD | 3.3 (3.6) | 2.9 (3.4) | 3.2 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate Per 100 Person Years of Hospitalization or Emergency Department (ED) Visit Related to Exacerbation of Chronic Obstructive Pulmonary Disease (COPD)
Description: A severe exacerbation is defined as one with a primary diagnosis of COPD. A moderate exacerbation is an ED visit with a primary diagnosis of COPD, a physician visit with a diagnosis of COPD and a prescription for an oral corticosteroid, a physician visit with a diagnosis code for COPD and an antibiotic for respiratory infection, or physician administration of nebulized albuterol within 3 days of an office visit. Incidence rate is calculated by dividing the number of exacerbations by the number of person years. Person years adjust for different lengths of follow up for participants.
Time Frame: Data were collected over a maximum period of 4 years
Population: Managed care enrollees (aged >40 years) with at least one COPD-related exacerbation at baseline and newly initiating therapy with TIO with or without the addition of FSC during the study enrollment period was the target population. The date of TIO-alone therapy or TIO+FSC add-on date was the index date.
Measure: Number; unit: exacerbations per 100 person years
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC)
Number analyzed (Participants) | 2481 | 852
exacerbations per 100 person years
  Any exacerbation | 95.58 | 75.38
  Severe exacerbation | 7.86 | 5.06
  Moderate exacerbation | 88.65 | 69.74
Statistical Analysis 1: Comparison: Tiotropium Bromide (TIO) vs TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC); Test type: Superiority or Other; p = 0.007, Regression, Logistic — COPD-Related Adjusted Multivariate Outcomes in the Follow-Up Period by Cohort (reference cohort = TIO) for Any COPD Exacerbation; Hazard Ratio (HR) = 0.772, 95% CI 2-sided [0.641 to 0.930]
Statistical Analysis 2: Comparison: Tiotropium Bromide (TIO) vs TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC); Test type: Superiority or Other; p = 0.146, Regression, Logistic — COPD-Related Adjusted Multivariate Outcomes in the Follow-Up Period by Cohort (reference cohort = TIO) for Severe COPD Exacerbations; Hazard Ratio (HR) = 0.622, 95% CI 2-sided [0.328 to 1.180]
Statistical Analysis 3: Comparison: Tiotropium Bromide (TIO) vs TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC); Test type: Superiority or Other; p = 0.013, Regression, Logistic — COPD-Related Adjusted Multivariate Outcomes in the Follow-Up Period by Cohort (reference cohort = TIO) for Moderate COPD Exacerbations; Hazard Ratio (HR) = 0.763, 95% CI 2-sided [0.646 to 0.949]

2. Secondary Outcome: Adjusted Mean Monthly Costs Per COPD Patient by Treatment Group
Description: The mean costs of health care encounters adjusted to control for baseline differences between treatment groups and reported in 2008 United States dollars as calculated with the consumer price index (CPI) are presented. CPI is standard multiplier for adjusting the cost of goods and services to a single year. Total costs include pharmacy and medical costs. Medical costs were computed from the paid amounts of medical claims with a primary diagnosis code for COPD. COPD-related pharmacy costs were computed from paid amounts of COPD-related prescription medications.
Time Frame: Data were collected over a maximum period of 4 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: United States dollars
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC)
Number analyzed (Participants) | 2481 | 852
United States dollars
  Total costs | 721 [190 to 2005] | 721 [149 to 2250]
  Pharmacy Costs | 190 [67 to 379] | 223 [62 to 490]
  Medical costs | 543 [66 to 3543] | 490 [42 to 4004]

3. Secondary Outcome: Incidence Rate of Hospitalizations and Emergency Room Visits Per 100 Person Years
Description: Unadjusted incidence rates per 100 person years of chronic obstructive pulmonary disease (COPD)-related hospitalizations and emergency department visits by treatment group are presented. Incidence rate is calculated by dividing the number of healthcare service encounters by the number of person years of follow up. Person years adjust for different lengths of follow up for individual participants
Time Frame: Data were collected over a maximum period of 4 years
Population: as for outcome 1
Measure: Number; unit: visits per 100 person years
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC)
Number analyzed (Participants) | 2481 | 852
visits per 100 person years
  COPD-related hospital and emergency room visits | 95.58 | 75.38
  Hospitalizations | 11.14 | 7.43
  Emergency department visits | 12.63 | 9.90

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Tiotropium Bromide (TIO) | TIO Plus FSC/Salmeterol Xinafoate in Combination (TIO + FSC)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.